CLINICAL TRIAL: NCT00104611
Title: A Randomized, Parallel-Group, Sham-Controlled, Multi-Center Study to Evaluate the Safety and Efficacy of the Neuronetics Model 2100 CRS Repetitive Transcranial Magnetic Stimulation (rTMS) System in Patients With Major Depression
Brief Title: Study of a Repetitive Transcranial Magnetic Stimulation (rTMS) Device for the Treatment of Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neuronetics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 44-01101-000
Record Dates: First submitted 2005-03-02; First posted 2005-03-03 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Repetitive Transcranial Magnetic Stimulation; rTMS; Non-invasive Neuromodulation; Antidepressant
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TMS (Active Comparator): Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment 5 days/week for up to 6 weeks
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Placebo (Placebo Comparator): Treatment 5 days/week for up to 6 weeks
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation

SUMMARY:
This trial will test the safety and efficacy of a rTMS device for the treatment of major depressive disorder (MDD). It is hypothesized that rTMS will have an antidepressant effect.

It is a 10-week, randomized, sham-controlled, multicenter trial in outpatients recruited in both academic and private research centers. It is comprised of three major phases: pre-study screening, acute treatment, and post-treatment taper. Eligible patients will be randomized to one of two rTMS treatment groups. One group will receive active rTMS treatment and one will receive an inactive, or sham, treatment. Each treatment takes about 45 minutes and is done on an outpatient basis. All trial related medical care is provided at no cost to the participant.

DETAILED DESCRIPTION:
This trial will test the safety and efficacy of a rTMS device for the treatment of major depressive disorder.

Major depression is one of the most prevalent and profoundly debilitating diseases worldwide. In a recent report, it is estimated that by the year 2020, depression will be second only to heart disease in magnitude of disease burden as determined by disability-adjusted life years.

Despite major advances in the treatment of depression in the last three decades, further improvements are needed. For instance, with respect to antidepressant pharmacotherapy, only 1/3 of patients are estimated to have a nearly full resolution of their clinical symptoms with their first medication trial. Indeed, partial remission or lack of response to treatment is experienced by the majority of patients. Even with serial trials of antidepressant medication, at least 10 to 15% of patients with major depression are estimated to experience limited benefit and remain chronically depressed with significant psychosocial morbidity. Some patients cannot tolerate the dosage and duration of antidepressant treatments required for treatment trials to be considered adequate. In such patients, intolerance of somatic treatments for major depression leads to chronicity and impaired function, and likely hinders long-term compliance with treatments. For many patients with treatment resistant depression (TRD), more complex regimens of polypharmacotherapy, or the use of electroconvulsive therapy (ECT) are the only currently available treatment options.

Repetitive transcranial magnetic stimulation (rTMS) is a promising alternative to treatments such as ECT or pharmacotherapy for patients presenting with MDD. An rTMS procedure is non-invasive, does not require anesthesia, and may be delivered in an appropriately staffed outpatient setting.

By creating a time-varying magnetic field that is unimpeded by the scalp and skull, TMS can focally and painlessly stimulate the cortex of awake individuals. Through the principle of magnetic induction, the localized pulsed magnetic field generated in the coil at the surface of the head induces an electrical current that depolarizes underlying superficial neurons. It is widely thought that rTMS produces its behavioral effects solely through the induction of current flow in cortex.

Several factors have driven the investigation of rTMS for the treatment of MDD. Early reports of changes in mood in normal participants, the non-invasive nature of rTMS, the favorable side effect profile compared to ECT, and the non-response of a number of MDD patients to pharmacotherapy and/or ECT, all have likely played a role. Since the initial studies, there has continued to be high interest in rTMS as an antidepressant treatment. Multiple trials have been conducted from researchers in diverse environments around the world. However, until now, there have been no rigorously conducted large, multicenter rTMS clinical trials in the treatment of patients with MDD. Because the published research has largely been conducted in single centers, the sample sizes in these antidepressant trials have been small. However, the majority of more than 20 reports have found modest to large antidepressant effects that increase over the trial period. By design, this trial will provide more robust information regarding the antidepressant effect of rTMS in the adult population of MDD patients.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis by DSM-IV criteria for Major Depressive Episode, single or recurrent episode as confirmed by the Structured Clinical Interview for the DSM-IV (SCID-IV), with the additional stipulation of a duration for this episode of greater than or equal to 4 weeks and CGI-S greater than or equal to 4
* Duration of current episode of depression less than 3 years (the definition of an episode is demarcated by a period of greater than or equal to 2 months when the patient did not meet full criteria for the DSM-IV definition of major depressive episode);
* Total HAM-D17 score of greater than or equal to 20 and Item 1 score greater than or equal to 2 at screening visit;
* Medication resistance to at least two different antidepressant treatments, defined as resistance to a minimum of 1 and a maximum of 4 antidepressant drug trials of adequate dose and duration in the current episode with adequate dose and duration defined as minimum level 3 on the Antidepressant Treatment History Form (ATHF); or, if patient has not received a sufficient number of antidepressant treatments to assess their medication resistance in the current episode, then the patient must meet level 3 medication resistance by ATHF criteria to at least 1 and no more than 4 drug trials in a previous episode.
* Patients who have not completed antidepressant trials of adequate dose and duration due to intolerance to therapy may be included if they have demonstrated intolerance to greater than or equal to 4 anti-depressant medications in the current or a previous episode, and did not meet ATHF criteria for a single adequate treatment trial in the current episode.
* Capable and willing to provide informed consent
* Signed HIPAA authorization
* Able to adhere with the treatment schedule, and withdrawal of ongoing pharmacotherapy
* If currently taking antidepressant pharmacotherapy, must be clinically appropriate to discontinue treatment with those agents.

Exclusion Criteria:

* Investigators, site personnel directly affiliated with this study, and their immediate families (immediate family is defined as a spouse, parent, child or sibling, whether by birth or legal adoption);
* Individuals diagnosed by the Investigator with the following conditions (current unless otherwise stated):

  * Depression secondary to a general medical condition, or substance-induced;
  * Seasonal pattern of depression as defined by DSM-IV
  * History of substance abuse or dependence within the past year (except nicotine and caffeine)
  * Any psychotic disorder (lifetime), including schizoaffective disorder, or major depression with psychotic features in this or previous episodes
  * Bipolar disorder
  * Eating disorder (current or within the past year)
  * Obsessive compulsive disorder (lifetime)
  * Post-traumatic stress disorder (current or within the past year)
* An Axis II Personality Disorder, which in the judgment of the Investigator may hinder the patient in completing the procedures required by the study protocol.
* Individuals with a clinically defined neurological disorder or insult including, but not limited to:

  * Any condition likely to be associated with increased intracranial pressure
  * Space occupying brain lesion
  * Any history of seizure EXCEPT those therapeutically induced by ECT
  * History of cerebrovascular accident
  * Transient ischemic attack within two years
  * Cerebral aneurysm
  * Dementia
  * Mini Mental Status Exam score of less than or equal to 24
  * Parkinson's disease
  * Huntington's chorea
  * Multiple sclerosis
* Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or history of significant head trauma with loss of consciousness for greater than or equal to 5 minutes
* A true positive response to any question on the Transcranial Magnetic Stimulation Adult Safety Screen questionnaire
* Inability to locate and quantify a motor threshold as defined in the protocol
* ECT treatment within 3 months prior to the screening visit
* Failure to respond to ECT treatment (i.e., consistent with ATHF level 2 or higher) in this or any previous episode
* History of treatment with rTMS therapy for any disorder
* History of treatment with Vagus Nerve Stimulation
* Use of any investigational drug within 4 weeks of the randomization visit
* Use of fluoxetine within 6 weeks of the randomization visit
* Use of an MAOI within 2 weeks of the randomization visit
* Use of any medication(s) listed on the Excluded Medication List within 1 week of the randomization visit
* Significant acute suicide risk, defined as follows:

  * Suicide attempt within the previous 6 months that required medical treatment; or
  * Greater than or equal to 2 suicide attempts in the past 12 months; or
  * Has a clear-cut plan for suicide and states that he/she cannot guarantee that he/she will call his/her regular psychiatrist or the Investigator if the impulse to implement the plan becomes substantial during the study; or
  * In the Investigator's opinion, is likely to attempt suicide within the next 6 months.
* Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease;
* Intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
* Known or suspected pregnancy
* If participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the rTMS trial
* Positive urine drug screen. (A positive urine drug screen at screening may be repeated once prior to randomization)
* Clinically significant laboratory abnormality, in the opinion of the Investigator
* Women who are breast-feeding
* Women of child-bearing potential not using a medically accepted form of contraception when engaging in sexual intercourse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2004-01; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
• Evaluate the antidepressant effect of a specified treatment course of rTMS compared to sham treatment given under the same experimental conditions | 4 to 6 weeks

SECONDARY OUTCOMES:
Safety and tolerability of rTMS | screening through 30 days past last day of participation
Change in depressive symptomatology with rTMS | acute phase
Short term durability of rTMS efficacy | during 3 week taper

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - PsyCare, Poway, California
  - Stanford University School of Medicine, Stanford, California
  - Northwestern University School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - UVA Center for Psychiatric Clinical Research, Charlottesville, Virginia

REFERENCES:
- [Derived] Janicak PG, Nahas Z, Lisanby SH, Solvason HB, Sampson SM, McDonald WM, Marangell LB, Rosenquist P, McCall WV, Kimball J, O'Reardon JP, Loo C, Husain MH, Krystal A, Gilmer W, Dowd SM, Demitrack MA, Schatzberg AF. Durability of clinical benefit with transcranial magnetic stimulation (TMS) in the treatment of pharmacoresistant major depression: assessment of relapse during a 6-month, multisite, open-label study. Brain Stimul. 2010 Oct;3(4):187-99. doi: 10.1016/j.brs.2010.07.003. Epub 2010 Aug 11. PMID 20965447
- [Derived] Demitrack MA, Thase ME. Clinical significance of transcranial magnetic stimulation (TMS) in the treatment of pharmacoresistant depression: synthesis of recent data. Psychopharmacol Bull. 2009;42(2):5-38. PMID 19629020
- [Derived] Simpson KN, Welch MJ, Kozel FA, Demitrack MA, Nahas Z. Cost-effectiveness of transcranial magnetic stimulation in the treatment of major depression: a health economics analysis. Adv Ther. 2009 Mar;26(3):346-68. doi: 10.1007/s12325-009-0013-x. Epub 2009 Mar 28. PMID 19330495
- [Derived] Avery DH, Isenberg KE, Sampson SM, Janicak PG, Lisanby SH, Maixner DF, Loo C, Thase ME, Demitrack MA, George MS. Transcranial magnetic stimulation in the acute treatment of major depressive disorder: clinical response in an open-label extension trial. J Clin Psychiatry. 2008 Mar;69(3):441-51. doi: 10.4088/jcp.v69n0315. PMID 18294022
- [Derived] Janicak PG, O'Reardon JP, Sampson SM, Husain MM, Lisanby SH, Rado JT, Heart KL, Demitrack MA. Transcranial magnetic stimulation in the treatment of major depressive disorder: a comprehensive summary of safety experience from acute exposure, extended exposure, and during reintroduction treatment. J Clin Psychiatry. 2008 Feb;69(2):222-32. doi: 10.4088/jcp.v69n0208. PMID 18232722
- [Derived] O'Reardon JP, Solvason HB, Janicak PG, Sampson S, Isenberg KE, Nahas Z, McDonald WM, Avery D, Fitzgerald PB, Loo C, Demitrack MA, George MS, Sackeim HA. Efficacy and safety of transcranial magnetic stimulation in the acute treatment of major depression: a multisite randomized controlled trial. Biol Psychiatry. 2007 Dec 1;62(11):1208-16. doi: 10.1016/j.biopsych.2007.01.018. Epub 2007 Jun 14. PMID 17573044